CLINICAL TRIAL: NCT02717650
Title: Development; Feasibility/Safety and Validation of the Alfred Step Test Exercise Protocol (A-STEP) Developed for Adults With Cystic Fibrosis:
Brief Title: The Alfred Step Test Exercise Protocol (A-STEP), for Adults With Cystic Fibrosis.
Acronym: A-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Lisa Wilson, Senior Physiotherapist, The Alfred
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: 205/16; 205/16 (Other: The Alfred Ethics Committee); 0267 (Other: Human Ethics Committee Monash University)
Record Dates: First submitted 2016-03-10; First posted 2016-03-24 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis; Fibrosis; Lung Diseases; Respiratory Diseases; Genetic Diseases; Pancreatic Diseases
Keywords: Exercise Testing; Maximal Exercise Testing; Maximal Exercise Capacity; Peak Exercise Capacity; Adults; Step Tests
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A-STEP (Experimental): Study A) A-STEP Study Development of new exercise test protocol and Observational Feasibility/Safety Study (no comparator).
  Interventions: Other: A-STEP
- A-STEP (New Protocol) (Experimental): Study B) A-STEPmax Study Validity Study (random allocation of test order).
  Interventions: Other: A-STEP (New Protocol)
- CPET cycle ergometer (Gold Standard) (Active Comparator): Study B) A-STEPmax Study Validity Study (random allocation of test order).
  Interventions: Other: Comparator: CPET cycle ergometer (Gold Standard)

INTERVENTIONS:
Other: A-STEP — Study A) Study A) Development of new exercise test protocol and Observational Feasibility/Safety Study (no comparator).
  Feasibility/safety of a newly designed, incremental, maximal, standardised step test in adults with Cystic Fibrosis.
  Other Names: Alfred Step Test Exercise Protocol (A-STEP)
  Arms: A-STEP
Other: A-STEP (New Protocol) — Study B) Validation Study (random allocation of test order). Validity of an incremental, maximal, standardised incremental step test with breath-by-breath gas analysis using portable metabolic measurement equipment against CPET.
  Other Names: Alfred Step Test Exercise Protocol
  Arms: A-STEP (New Protocol)
Other: Comparator: CPET cycle ergometer (Gold Standard) — Study B) Validation study (random allocation of test order) "Gold standard" CPET. An incremental, maximal standardised cycle ergometer exercise test (performed as per published protocol) using portable metabolic measurement equipment.
  Other Names: Cardiopulmonary Exercise Test Protocol
  Arms: CPET cycle ergometer (Gold Standard)

SUMMARY:
Exercise testing has become clinically important in the management and ongoing evaluation of patients with Cystic Fibrosis (CF) with higher rates of exercise tolerance and participation previously linked to lower mortality risk (1).

Lower exercise capacity generally correlates with more severe lung disease (2,3) and landmark studies suggest that low exercise capacity as measured by peak oxygen capacity (VO2peak) and rate of decline in lung function (FEV1) are strong predictors of mortality (1,4). However not all studies have found pulmonary function tests (PFTs) to be reliable predictors of maximal exercise capacity (5), especially in relatively well preserved lung function (6,7).

The wide distribution in physical capacity between fit individuals and end stage disease adds to complexity of assessment. Independent factors of age, genetics, habitual exercise, nutritional status and musculoskeletal conditions are all known to influence physical capacity in patients with CF (8,9).

Maximal exercise testing places additional stress on cardiovascular, respiratory and peripheral systems providing more information around multiple influences on disease progression including degree of limitation in these major systems (10,11) and is useful for assessment of exercise desaturation, more common (but not always present) in advanced lung disease (5,12).

With prediction of exercise performance and functional capacity from PFTs unreliable and the understanding that health status correlates better with exercise tolerance there has been an increase in maximal exercise testing for patient management (13). Many international centers now regard exercise testing as highly important with many assessing maximal exercise capacity annually to monitor disease progression, identify physical status and drive changes in medical, physiotherapy or nutritional management (14,15).

The main vision is to develop a standardized incremental step test protocol suitable for adults with Cystic Fibrosis (CF), all ages, levels of fitness and disease state that is in line with current exercise testing recommendations (15). To develop a more useful field test to assess exercise tolerance and a more "user friendly" test than the currently available laboratory exercise test to allow for early detection of decline in physical function in the day-to-day clinical setting. To date no studies have been published in adults with CF where an incremental exercise step test has been investigated to assess exercise tolerance or determine maximum oxygen uptake (VO2max).

DETAILED DESCRIPTION:
Many international centers now regard exercise testing as highly important with many measuring maximal exercise capacity annually to monitor disease progression, identify physical status and to drive changes in medical, physiotherapy or nutritional management (14,15).

Cardiopulmonary Exercise Testing (CPET):

The current best practice for assessing VO2max in adults with CF is a CPET using the Godfrey Protocol, a progressive and incremental maximal test performed on a cycle ergometer (13,14,15). Exercise testing should aim to achieve a maximal response within a time frame of 8-12 min and incremental protocols with stage duration of 1 minute are considered more efficient in eliciting the desired response within this time frame (14). During CPET, VO2max is determined while breath-by-breath gas analysis allows for a comprehensive assessment of exercise ventilation and circulation. This information can identify reasons for low exercise capacity and whether exercise limitation is due to deconditioning, or primarily within the respiratory, cardiovascular or peripheral systems. CPET is performed using a specialist ergometer, and requires specialist clinical expertise, monitoring and reporting equipment for interpretation of the test. The cost, space and expertise to carry out CPET in CF units around the world may limit its use for the regular assessment of exercise capacity in adults with CF (16).

Field Tests:

Field tests generally cannot determine absolute maximal exercise capacity, but do provide valuable information about the patient's functional abilities and limitations and compared to laboratory tests are inexpensive and easy to administer.

Field tests that use a single step for assessment of exercise tolerance in patients with chronic lung disease include:

3-Minute Step Test (3MST):

The 3MST is a feasible and acceptable measure of sub-maximal exercise performance in children and adults and a useful tool in the assessment of oxygen desaturation (17,18). The test is short in duration, simple to carry out, and has low cost and minimal space and equipment requirements however the sub-maximal nature and ceiling effect of the 3MST limits its usefulness clinically across the age spectrum (18,19).

The Chester Step Test (CST):

The CST is a 10-minute sub-maximal standardized multistage test and like the 3MST has minimal space and equipment requirements. The CST was originally designed for workplace screening and is now widely used for exercise prescription in the UK cardiac population (20). In healthy individuals one study reported a ceiling effect and a positive relationship between predicted VO2max using the CST and measured VO2max (21) however a subsequent study questioned this prediction validity (22). The CST has been found to be highly reproducible in patients with chronic obstructive lung disease (COPD) and reliable in patients with Bronchiectasis, but too challenging for both groups (23,24).

The Modified Incremental Step Test (MIST):

The MIST was designed to be more suitable for COPD patients and modeled from the CST(25). A reduction in work rate was not found to result in a difference in cardiopulmonary stress and exertion effort at peak exercise but did result in a higher exercise tolerance in patients with COPD. The MIST is reliable and better tolerated than the CST in patients with Bronchiectasis (23,24).

The CST and CF:

One study (published in abstract form) has shown the CST to be a useful field test when compared to the 3MST and 6MWT for those with mild to moderate CF. The authors commented this was likely due to the progressive nature being more representative of adult physical activity (26).

The main vision is to develop a standardized incremental step test protocol suitable for adults with Cystic Fibrosis (CF), all ages, levels of fitness and disease state that is in line with current exercise testing recommendations (15). The test should be a more useful than the already available field tests and more "user friendly" test than the currently available laboratory exercise test to assess exercise tolerance and allow for early detection of decline in physical function in the day-to-day clinical setting. To date no studies have been published in adults with CF where an incremental exercise step test has been investigated to assess exercise tolerance or determine VO2max.

1. To design a standardized externally paced incremental step test that is portable, easy to administer, simple to perform, time, cost and space efficient (A-STEP).

   Study A:
2. To assess feasibility and reliability of the A-STEP to objectively assess exercise tolerance.
3. To determine if the A-STEP is a more useful tool than the 3-Minute Step Test.

   Study B:
4. To develop an alternative tool to determine maximum oxygen uptake (VO2max) to the "gold standard" CPET that is feasible across the whole spectrum of lung disease.
5. To determine if the A-STEPmax is a valid tool when compared to the VO2max achieved from a CPET performed on a cycle ergometer using the Godfrey Protocol.

The principle investigator hypothesizes that the A-STEP will be a feasible tool to assess exercise capacity; and the A-STEP max will be a valid tool for the assessment of VO2max across the age range and disease spectrum in adults with CF.

ELIGIBILITY:
INCLUSION

* Confirmed Diagnosis of CF (by genotype or positive sweat test)
* Aged 18yrs and older
* FEV1 ≥20% (Forced expiration in 1 sec)
* Stable baseline state. (Stable baseline state is defined as: clinically stable respiratory status, for at least 30 days, characterized by the absence of hospitalization and no changes in maintenance therapy during this period (Yankaskas et al 2004)).

EXCLUSION

* Febrile
* Haemoptysis
* Uncontrolled asthma
* Pneumothorax
* Cardiac issues
* Unreliable readings on pulse oximetry
* Pulmonary hypertension
* Unstable CF related diabetes (CFRD)
* Vascular issues
* Renal disease
* Pregnancy
* Body mass index (BMI) <18.0
* Significant musculoskeletal issues
* Unable to safely follow instructions

(ATS/ACCP 2003; Hebestreit 2015)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Study B) Maximum oxygen uptake (VO2max) | Measured during the incremental test for a maximum of 15 minutes.
  The highest oxygen uptake achieved during the exercise test taken from inspired gas in a given period of time. Body weight is used to calculate this from oxygen consumption during the test. VO2peak may be used as a surrogate if VO2max is not achieved. Criteria for reaching maximum effort is not included in this document.
Study A) Oxygen Saturation | Measured for 3 min prior to exercise (recorded at baseline sitting and standing), monitored during the test (recorded at minute intervals) and for at least 2 min of recovery up to a maximum of 10 minutes.
  Standard objective outcome measures of field exercise testing. Measured via pulse oximetry.
Study A) Heart Rate | Measures for 3 min prior to exercise (recorded at baseline sitting and standing), monitored during the test (recorded at minute intervals) and for at least 2 min of recovery up to a maximum of 10 minutes.
  Standard objective outcome measures of field exercise testing. Measured via pulse oximetry.

SECONDARY OUTCOMES:
Study B) Carbon Dioxide Production | Measured during the test incremental tests for a maximum 15 minutes and 5 mins of recovery.
  Standard secondary outcome measure of maximal exercise testing using breath- by-breath gas analysis with portable metabolic measurement equipment.
Study B) Respiratory Exchange Ratio | Measured during the test incremental tests for a maximum 15 minutes and 5 mins of recovery.
  Standard secondary outcome measure of maximal exercise testing using breath- by-breath gas analysis. The ratio of carbon dioxide production to oxygen consumption.
Study B) Minute Ventilation | Measured during the test incremental tests for a maximum 15 minutes and 5 mins of recovery.
  Standard secondary outcome measure of maximal exercise testing using breath- by-breath gas analysis. The product of tidal volume and respiratory rate.
Study B) Oxygen Pulse | Measured during the test incremental tests for a maximum 15 minutes and 5 mins of recovery.
  Standard secondary outcome measure of maximal exercise testing using breath- by-breath gas analysis. Calculated by dividing the oxygen consumption by heart rate.
Study B) Tidal Volume | Measured during the test incremental tests for a maximum 15 minutes and 5 mins of recovery.
  Standard secondary outcome measure of maximal exercise testing using breath- by-breath gas analysis. The volume of each breath taken.
Study B) Oxygen Saturation | easures are taken at baseline (post 5 mins), monitored during the test (recorded at minute intervals) and for min 5 mins of recovery
  Standard objective outcome measures of exercise testing. Measured via pulse oximetry.
Study B) Heart rate | easures are taken at baseline (post 5 mins), monitored during the test (recorded at minute intervals) and for min 5 mins of recovery
  Standard objective outcome measures of exercise testing. Measured via pulse oximetry.
Study B) Measures from Electrocardiogram | easures are taken at baseline (post 5 mins), monitored during the test (recorded at minute intervals) and for min 5 mins of recovery
  Used to monitor the patient's cardiac rhythm (CPET only)
Study A & B) Breathlessness and Leg Fatigue | Measures are taken at baseline (post 5 mins), monitored during the test (recorded at minute intervals) and for min 5 mins of recovery
  Standard subjective outcome measures of exercise testing. Modified Borg 0-10.
Study A & B) Blood pressure | Measures are takenpre/post A-STEP, pre/every 2 mins during/post CPET
  Standard outcome measure of exercise testing.
Study A & B) Duration of test; Highest level (mins and sec)/stage achieved; Reason for test termination. | Measured during or on completion of the test. Maximum 15 minutes.
  Parameters of exercise test.

OTHER OUTCOMES:
Study A & B) Gender; Age, Height, BMI, fitness level | Recorded on the day of testing maximum 10 mins.
  Demographic baseline descriptive measures.
Study A & B) Spirometry (Pulmonary Function Tests) | Recorded on the day of testing prior to testing, maximum 10 minutes Study B. Most recent PFTs if day of testing lung function is not available study A.
  Baseline Pulmonary Function Test measures.
Study A & B) Alfred Wellness Score for CF (AweScore CF) | Recorded on the day of testing prior to testing, maximum 2 minutes.
  Alfred specific clinical tools: quality of life measure.
Study A) Musculoskeletal Assessment Tool-Quick Screen | Recorded on the day of testing, maximum 20 minutes.
  Alfred specific clinical tool: to screen for musculoskeletal issues.
Study A & B) Medical history. | Recorded on the day of testing, maximum 10 minutes.
  Baseline descriptive measures of health status.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wilson, BHS(Physio), Principal Investigator — Alfred Hospital; Monash University
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data.

REFERENCES:
- [Background] Nixon PA, Orenstein DM, Kelsey SF, Doershuk CF. The prognostic value of exercise testing in patients with cystic fibrosis. N Engl J Med. 1992 Dec 17;327(25):1785-8. doi: 10.1056/NEJM199212173272504. PMID 1435933
- [Background] Godfrey S, Mearns M. Pulmonary function and response to exercise in cystic fibrosis. Arch Dis Child. 1971 Apr;46(246):144-51. doi: 10.1136/adc.46.246.144. PMID 5576246
- [Background] Marcotte JE, Grisdale RK, Levison H, Coates AL, Canny GJ. Multiple factors limit exercise capacity in cystic fibrosis. Pediatr Pulmonol. 1986 Sep-Oct;2(5):274-81. doi: 10.1002/ppul.1950020505. PMID 3774384
- [Background] Pianosi P, Leblanc J, Almudevar A. Peak oxygen uptake and mortality in children with cystic fibrosis. Thorax. 2005 Jan;60(1):50-4. doi: 10.1136/thx.2003.008102. PMID 15618583
- [Background] Henke KG, Orenstein DM. Oxygen saturation during exercise in cystic fibrosis. Am Rev Respir Dis. 1984 May;129(5):708-11. doi: 10.1164/arrd.1984.129.5.708. PMID 6426354
- [Background] Moorcroft AJ, Dodd ME, Webb AK. Exercise testing and prognosis in adult cystic fibrosis. Thorax. 1997 Mar;52(3):291-3. doi: 10.1136/thx.52.3.291. PMID 9093351
- [Background] Shah AR, Gozal D, Keens TG. Determinants of aerobic and anaerobic exercise performance in cystic fibrosis. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1145-50. doi: 10.1164/ajrccm.157.4.9705023. PMID 9563732
- [Background] Lands LC, Heigenhauser GJ, Jones NL. Respiratory and peripheral muscle function in cystic fibrosis. Am Rev Respir Dis. 1993 Apr;147(4):865-9. doi: 10.1164/ajrccm/147.4.865. PMID 8466121
- [Background] Nixon PA, Orenstein DM, Kelsey SF. Habitual physical activity in children and adolescents with cystic fibrosis. Med Sci Sports Exerc. 2001 Jan;33(1):30-5. doi: 10.1097/00005768-200101000-00006. PMID 11194108
- [Background] Barry SC, Gallagher CG. Corticosteroids and skeletal muscle function in cystic fibrosis. J Appl Physiol (1985). 2003 Oct;95(4):1379-84. doi: 10.1152/japplphysiol.00506.2002. Epub 2003 Jun 13. PMID 12807896
- [Background] Urquhart DS. Exercise testing in cystic fibrosis: why (and how)? J R Soc Med. 2011 Jul;104 Suppl 1(Suppl 1):S6-14. doi: 10.1258/jrsm.2011.s11102. No abstract available. PMID 21719895
- [Background] Rogers D, Prasad SA, Doull I. Exercise testing in children with cystic fibrosis. J R Soc Med. 2003;96 Suppl 43(Suppl 43):23-9. No abstract available. PMID 12906322
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Hebestreit H, Arets HGM, Aurora P, Boas S, Cerny F, Hulzebos EHJ, Karila C, Lands LC, Lowman JD, Swisher A, Urquhart DS; European Cystic Fibrosis Exercise Working Group. Statement on Exercise Testing in Cystic Fibrosis. Respiration. 2015;90(4):332-351. doi: 10.1159/000439057. Epub 2015 Sep 9. PMID 26352941
- [Background] Stevens D, Oades PJ, Armstrong N, Williams CA. A survey of exercise testing and training in UK cystic fibrosis clinics. J Cyst Fibros. 2010 Sep;9(5):302-6. doi: 10.1016/j.jcf.2010.03.004. Epub 2010 Mar 31. PMID 20359963
- [Background] Balfour-Lynn IM, Prasad SA, Laverty A, Whitehead BF, Dinwiddie R. A step in the right direction: assessing exercise tolerance in cystic fibrosis. Pediatr Pulmonol. 1998 Apr;25(4):278-84. doi: 10.1002/(sici)1099-0496(199804)25:43.0.co;2-g. PMID 9590488
- [Background] Holland AE, Rasekaba T, Wilson JW, Button BM. Desaturation during the 3-minute step test predicts impaired 12-month outcomes in adult patients with cystic fibrosis. Respir Care. 2011 Aug;56(8):1137-42. doi: 10.4187/respcare.01016. Epub 2011 Apr 15. PMID 21496365
- [Background] Narang I, Pike S, Rosenthal M, Balfour-Lynn IM, Bush A. Three-minute step test to assess exercise capacity in children with cystic fibrosis with mild lung disease. Pediatr Pulmonol. 2003 Feb;35(2):108-13. doi: 10.1002/ppul.10213. PMID 12526071
- [Background] Andrade CH, Cianci RG, Malaguti C, Corso SD. The use of step tests for the assessment of exercise capacity in healthy subjects and in patients with chronic lung disease. J Bras Pneumol. 2012 Jan-Feb;38(1):116-24. doi: 10.1590/s1806-37132012000100016. English, Portuguese. PMID 22407048
- [Background] Sykes, K., Roberts, A. . (2004). The Chester step test-a simple yet effective tool for the prediction of aerobic capacity. Physiotherapy Theory & Practice, 90(4 ), 183-188 doi: DOI: 10.1016/j.physio.2004.03.008)
- [Background] Buckley JP, Sim J, Eston RG, Hession R, Fox R. Reliability and validity of measures taken during the Chester step test to predict aerobic power and to prescribe aerobic exercise. Br J Sports Med. 2004 Apr;38(2):197-205. doi: 10.1136/bjsm.2003.005389. PMID 15039259
- [Background] de Camargo AA, Justino T, de Andrade CH, Malaguti C, Dal Corso S. Chester step test in patients with COPD: reliability and correlation with pulmonary function test results. Respir Care. 2011 Jul;56(7):995-1001. doi: 10.4187/respcare.01047. PMID 21740727
- [Background] Camargo AA, Lanza FC, Tupinamba T, Corso SD. Reproducibility of step tests in patients with bronchiectasis. Braz J Phys Ther. 2013 May-Jun;17(3):255-62. doi: 10.1590/s1413-35552012005000089. PMID 23966142
- [Background] de Andrade CH, de Camargo AA, de Castro BP, Malaguti C, Dal Corso S. Comparison of cardiopulmonary responses during 2 incremental step tests in subjects with COPD. Respir Care. 2012 Nov;57(11):1920-6. doi: 10.4187/respcare.01742. Epub 2012 Jun 15. PMID 22709990
- [Background] Planner, S., Morrison, L., Campbell, J., Bicknell, S., Ross, E. (2007). The Chester Step Test-Is this a Valid Predictor of Disease Severity in Adult CF? . Paper presented at the 2007 Cystic Fibrosis Conference.
- [Background] Wilson LM, Ellis MJ, Lane RL, Wilson JW, Keating DT, Jaberzadeh S, Button BM. Development of the A-STEP: A new incremental maximal exercise capacity step test in cystic fibrosis. Pediatr Pulmonol. 2021 Dec;56(12):3777-3784. doi: 10.1002/ppul.25667. Epub 2021 Sep 17. PMID 34499432